CLINICAL TRIAL: NCT04481945
Title: Evaluation of Antimicrobial Efficacy and Adaptability to Root Canal Dentin of Bioceramic Sealer Containing Nanoparticles (In-vitro Study)
Brief Title: Evaluation of Antimicrobial Efficacy and Adaptability of Bioceramic Sealer Containing Nanoparticles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Nourhan Magdy Yehia, Principal investigator, Misr International University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: END 6115018
Record Dates: First submitted 2019-06-25; First posted 2020-07-22 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: Nanosilver and chitosan inserted to BC sealer and so the antibacterial activity will be assessed on E. faecalis using direct contact test after the setting of the sealer, and the results will be reported using percentage reduction of the colony forming units.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding; Assessor blinding, where both the evaluators and statisticians will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- bioceramic sealer (Active Comparator): pre-mixed bioceramic obturation material. It is dispensed using a syringe in cases of root canal obturation and with either a syringe or as a putty when doing root repair and retrograde fillings.
  Interventions: Drug: bioceramic sealer
- bioceramic sealer and silver nanoparticles (Experimental): silver nanoparticles are antibacterial ions that can interact with multiple targets in the bacterial cell
  Interventions: Drug: bioceramic sealer
- bioceramic sealer and chitosan (Experimental): chitosan has an excellent antibacterial, antiviral and antifungal properties, as an antibacterial, it works better on gram negative than gram positive
  Interventions: Drug: bioceramic sealer

INTERVENTIONS:
Drug: bioceramic sealer — pre-mixed bioceramic obturation material. It is dispensed using a syringe in cases of root canal obturation and with either a syringe or as a putty when doing root repair and retrograde fillings.
  Other Names: total fill

SUMMARY:
Successful endodontic treatment depends primarily on the elimination of infecting microorganisms. This is done by chemo-mechanical preparation of root canals, which is not enough and microorganisms might still survive. Thus, from the main requirements of sealers is to have antibacterial properties and adaptability. Those requirements are needed to kill persisting bacteria after obturation and provide effective seal. Therefore, nanosilver and chitosan inserted to BC sealer and so the antibacterial activity will be assessed on E. faecalis using direct contact test after the setting of the sealer, and the results will be reported using percentage reduction of the colony forming units. Besides, adaptability will be assessed using scanning electron microscope.

DETAILED DESCRIPTION:
The main purpose of endodontic therapy is to clean and shape the root canals. This is done by means of instruments and chemical irrigants in order to effectively control the pulpal and periapical infection. That chemomechanical preparation aims to reduce the microorganisms count but cannot completely eliminate it. This is mainly due to (i) anatomical complexity and access limitations (ii) incompetent chemomechanical preparations leaving surfaces untouched (iii) ineffectual irrigation. Besides, despite an accurate chemomechanical preparation, infection may persist in 20-33% of cases, even if intracanal medicament is used.

Treatment failure may also occur due to microleakage, which occurs due to interfacial gaps between the gutta-percha and the sealer, the sealer and the dentin, or through voids within the sealer. Fifty eight percent of treatment failures happen due to incomplete obturation and that's why, hermetic seal is the main factor associated with the success of root canal treatment . Therefore, disinfection, gap-free, three dimensional obturation are the main requisites for treatment standards in endodontics.

Another reason for treatment failure is presence of persisting bacteria. Enterococcus faecalis is a resistant bacterium commonly retrieved from obturated root canals with post treatment disease (apical periodontitis). This pathogen is believed to be highly virulent; it can invade dentinal tubules, adhere, overcome environmental challenges and form biofilm.. Besides, it can resist intracanal disinfectants and medicaments. Therefore, the best approach to resolve this is by using a sealer with broad spectrum antibacterial action.

Ideal root-canal sealer should be able to kill microorganisms on direct contact on the dentinal walls and those present deep inside the dentinal root canals. That means that it should be able to diffuse inside the dentinal tubules to entomb and kill surviving bacteria. Besides, it should be capable of perfectly sealing the prepared canal to block any space and nutrients needed for bacterial growth. Finally, endodontic sealers that retain flowability and antimicrobial properties may help eliminate microorganisms in the root canal system.

Dspite the fact that most sealers have antibacterial constituents, their antibacterial activity is eventually lost after setting. Besides, even if it doesn't, these constituents have to be liberated from the set sealer matrix to fulfill their function. Then again, their release would be accompanied by disintegration of the sealer, interfacial gaps and later on bacterial recolonization.

Moreover,the current root filling materials aren't enough for reaching a complete, gap-free obturation. That would be due to the dimensional changes and lack of adhesion between Gutta percha and dentin. And that is why endodontic sealers are used. Thus, the adaptability of the sealer to the dentin is the main factor influencing microleakage and reinfection.

Nanotechnology is the science of producing materials in nano-dimensions by re-location and re-arrangement of atoms to prepare materials with better properties. It is considered a great advancement in the field of medicine. It can be beneficial in producing material with superior properties by enhancing surface to volume ratio. Besides, having antibacterial nanoparticles are shown to have better antibacterial action than their powder counterparts. That would be due to their higher surface area and charge density which favor their interaction with the negatively charged bacterial surface.

Resistance in pathogens is a major challenge in field like biomedicine. Chemical antimicrobial agents depend on binding to specific receptor for their antimicrobial action, which by time lead to multidrug resistance. . On the other hand, antibacterial nanoparticles such as nanosilver interact with multiple targets in the bacterial cell. Therefore, providing the bacteria with the least chance of gaining resistance.

The mechanism of action of silver ions. Silver ions are highly reactive. They start by binding to proteins on the bacterial cell leading to structural changes, which leads to cell distortion and death. Silver ions also can inhibit the bacterial replication, by binding and denaturing its DNA. Moreover, they can react with thiol group of proteins, followed by DNA condensation resulting in the cell death.

Although, silver nanoparticle's potential disadvantage is its toxicity towards mammalian cells. A number of studies proved that silver is safe as long as it's used in small concentrations. A study assessed the tissue response of silver nanoparticles dispersion embedded in fibrin sponge and implanted in polyethylene tubes. They concluded that silver nanoparticles dispersion was biocompatible at low concentrations. Another study stated that silver nanoparticles at low concentrations are effective against microorganisms without any toxic effect on eukaryotic cells.

Furthermore, there is a natural cationic biopolymer which can overcome the silver nanoparticles shortcomings and still provide an antibacterial efficacy. Chitosan (CS) is usually obtained by the alkaline deacetylation of chitin, which is the main component of the exoskeleton of crustaceans. CS has an excellent antibacterial, antiviral and antifungal properties, as an antibacterial, it works better on gram negative than gram positive. Besides, the addition of CS nanoparticles into zinc-oxide eugenol sealer in a membrane restricted assay. They proved that CS improved the antibacterial property suggesting that it can diffuse and penetrate dentinal tubules and anatomical complexities.

The mechanism of action of CS and stated that it's contact-mediated killing. It starts by electrostatic attraction of positively charged CS with negatively charged bacterial cell membrane. That is followed by altered cell permeability, resulting in rupture of cells and leakage of the intracellular components.

Finally, as reflected earlier, successful endodontic treatment depend on disinfecting the canals and providing a hermetic seal. That's why; this study's target is to assess the antibacterial efficacy and adaptability of bioceramic sealer when incorporated with nanosilver and chitosan respectively.

ELIGIBILITY:
Inclusion Criteria:

* Sound extracted anterior without any signs of caries
* No cracks
* No resorption or immature apices
* Single rooted with single canal confirmed radiographically both buccolingually and mesiodistally

Exclusion Criteria:

* Calcified canals
* Internal or external resorption
* Crown or root fractures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Antibacterial efficacy Measuring antibacterial effect of sealers | 24 hours
  Counting the colony forming units (in-vitro study)

SECONDARY OUTCOMES:
adaptability | 24 hours
  Assessment of adaptation using scanning electron microscope

CONTACTS AND LOCATIONS:
Overall Officials: N M Yehia, MA, Principal Investigator — teaching assistant at Misr International University
Locations (1):
- Misr International university, Faculty of Oral and Dental Medicine, Cairo, Egypt

REFERENCES:
- [Background] 1. Ricucci D, Siqueira JF. Fate of the Tissue in Lateral Canals and Apical Ramifications in Response to Pathologic Conditions and Treatment Procedures. Journal of Endodontics. 2010;836(1):1-15. 2. Waltimo T, Trope M, Haapasalo M, Ørstavik D. Clinical efficacy of treatment procedures in endodontic infection control and one year follow-up of periapical healing. J Endod. 2005;31(12):863-66. 3. Khayat A, Lee SJ, Torabinejad M. Human saliva penetration of coronally unsealed obturated root canals. J Endod. 1993 ;19(9):458-61. 4. Ingle J, Bakland L, Baumgartner J. Endodontics 6. 2008. 997-1018 p. 5. Kayaoglu G, Erten H, Alaçam T, Ørstavik D. Short-term antibacterial activity of root canal sealers towards Enterococcus faecalis. Int Endod J. 2005;38(7):483-88. 6. Wu D, Fan W, Kishen A, Gutmann JL, Fan B. Evaluation of the antibacterial efficacy of silver nanoparticles against Enterococcus faecalis biofilm. J Endod [Internet]. 2014;40(2):285-90. 7. Alabdulmohsen ZA, Saad AY. Antibacterial effect of silver nanoparticles against Enterococcus faecalis. Saudi Endod J. 2017;7(1):29-35. 8. Monajemzadeh A, Ahmadi Asoor S, Aslani S, Sadeghi-Nejad B. In vitro antimicrobial effect of different root canal sealers against oral pathogens. Curr Med Mycol. 2017; 3(2):7-12. 9. Barros J, Silva MG, Rodrigues MA, Alves FRF, Lopes MA, Pina-Vaz I, et al. Antibacterial, physicochemical and mechanical properties of endodontic sealers containing quaternary ammonium polyethylenimine nanoparticles. Int Endod J. 2014;47(8):725-34. 10. ElKateb WM, Massoud AG, Mokhless NA, Shalaby TI. Measurement of Tubular Penetration Depth of Three Types of Nanoparticles Mixed With Endodontic Sealer Using Scanning Electron Microscope (An in vitro study). J Am Sci. 2015;11(11):111-22. 11. HUANG Y, ORHAN K, CELIKTEN B, ORHAN AI, TUFENKCI P, SEVIMAY S. Evaluation of the sealing ability of different root canal sealers: a combined SEM and micro-CT study. J Appl Oral Sci [Internet]. 2018;26(0):1-8. 12. Naghavi N, Mortazavi M, Nejat A, Javidi M, Zarei M. Zinc oxide nano-particles as sealer in endodontics and its sealing ability. Contemp Clin Dent. 2014; Jan-Mar;5(1):20-24. 13. Kim JS, Kuk E, Yu KN, Kim JH, Park SJ, Lee HJ, et al. Antimicrobial effects of silver nanoparticles. Nanomedicine Nanotechnology, Biol Med. 2007;3(1):95-101. 14. Rai MK, Deshmukh SD, Ingle AP, Gade AK. Silver nanoparticles: The powerful nanoweapon against multidrug-resistant bacteria. J Appl Microbiol. 2012;112(5):841-52. 15. Gomes-Filho JE, Silva FO, Watanabe S, Angelo Cintra LT, Tendoro KV, Dalto LG, et al. Tissue Reaction to Silver Nanoparticles Dispersion as an Alternative Irrigating Solution. J Endod [Internet]. 2010 Oct 1;36(10):1698-702. 16. Kangarlou A, Tashfam B, Naseri M, Dianat O, Taheri S. In Vitro Comparison of Antibacterial Efficacy of a New Irrigation Solution Containing Nanosilver with Sodium Hypochlorite and Chlorhexidine. J Dent Sch. 2013;31(1):1-7. 17. Del Carpio-Perochena A, Kishen A, Shrestha A, Bramante CM. Antibacterial Properties Associated with Chitosan Nanoparticle Treatment on Root Dentin and 2 Types of Endodontic Sealers. J Endod. 2015; 41(8):1353-58. 18. Rabea EI, Badawy MET, Stevens C V., Smagghe G, Steurbaut W. Chitosan as antimicrobial agent: Applications and mode of action. Vol. 4, Biomacromolecules. 2003. p. 1457-65. 19. Kishen A, Shi Z, Shrestha A, Neoh KG. An Investigation on the Antibacterial and Antibiofilm Efficacy of Cationic Nanoparticulates for Root Canal Disinfection. J Endod. 2008;34(12):1515-20 20. Shrestha A, Kishen A. Antibacterial Nanoparticles in Endodontics: A Review. J Endod. 2016;42(10):1417-26. 21. Wang Z, Shen Y, Haapasalo M. Dentin extends the antibacterial effect of endodontic sealers against Enterococcus faecalis biofilms. J Endod. 2014;40(4):505-8.